CLINICAL TRIAL: NCT06934525
Title: Testing Delivery of Modalities in Community Health Settings: Developing Pathways to Health Equity
Brief Title: Implementing Team-Based Treatment for Pediatric Anxiety in Community Mental Health Settings
Acronym: IMPACT-RI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPS2023C233953
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-04

CONDITIONS: Obsessive Compulsive Disorder (OCD); Pediatric Anxiety Disorders; Anxiety Disorder; Anxiety; OCD; Phobia; Agoraphobia; Generalized Anxiety; Generalized Anxiety Disorder; Selective Mutism; Separation Anxiety; Social Anxiety; Social Anxiety Disorder; Panic Disorder; Pediatric Disorders
Keywords: exposure therapy; cognitive behavioral therapy; anxiety treatment; exposure and response prevention therapy; ERP; pediatric anxiety treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Phobic Disorders; Agoraphobia; Generalized Anxiety Disorder; Mutism; Anxiety, Separation; Phobia, Social; Panic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flexible (Other): Families and providers will collaboratively choose treatment delivery modality (in-person versus telehealth) on a session-by-session basis.
  Interventions: Behavioral: Team-delivered, exposure-based CBT
- In-person (Other): Families will only attend sessions in-person. Sessions may occur at the family's home, in the community, or in the provider's office.
  Interventions: Behavioral: Team-delivered, exposure-based CBT
- Telehealth (Other): Families will only attend sessions via a secure remote video platform.
  Interventions: Behavioral: Team-delivered, exposure-based CBT

INTERVENTIONS:
Behavioral: Team-delivered, exposure-based CBT — Patient sees licensed provider 1x/month and non-licensed provider 3x/month for exposure-based cognitive behavioral therapy

SUMMARY:
The purpose of this study is to test how the delivery of Cognitive Behavioral Therapy (CBT) for pediatric anxiety and OCD via different methods might increase its availability and effectiveness. CBT involves teaching the patient skills to enable them to gradually come into contact with feared situations. This process of gradually approaching feared situations is called exposure. Although CBT with exposure has the best evidence for treating anxiety disorders, not all children have equal access or respond the same way to CBT. As part of this study, patients will receive weekly CBT treatment sessions involving a combination of weekly visits with an exposure coach and one visit a month with a licensed provider (e.g., psychologist, social worker). This treatment will be delivered using one of three methods: 1) in-person (face-to-face sessions, occurring in the office and the home/community), or 2) telehealth (entirely remote sessions via web-based video conference), or 3) flexible (individualized mix of in-person and/or telehealth sessions). Eligible participants will be randomly assigned to one of these three methods. Results of this study will help determine which treatment method works best for whom.

Treatment as described above will occur as part of care at partnering community care sites in Rhode Island. Providers from the following partnering community care sites will make up patient treatment teams: Blackstone Valley Community Health Care, Family Services of Rhode Island, Gateway Healthcare, Newport Mental Health, and Thrive Behavioral Health.

The research study is being conducted by the Pediatric Anxiety Research Center at Brown University Health. The research team will conduct the study assessments that patients will be asked to participate in as study participants. Patients will be asked to complete assessments prior to starting treatment, at two time points during treatment, at the end of treatment, and at two timepoints 3 and 6 months following the end of treatment. Participants will be compensated for their time completing research assessments.

DETAILED DESCRIPTION:
The goal of this study is to increase equitable access to high quality care for all youth with anxiety and their families by comparing treatment modalities to determine which is best for whom in a comprehensive, state-wide approach (Rhode Island; RI) involving collaboration with a robust partner network offering a wide range of relevant experiences and expertise. To deliver care, the study team is partnering with Certified Community Behavioral Health Centers and a Federally Qualified Health Center representing a large proportion of historically marginalized youth across RI. Study results will inform the optimal delivery modality for enabling organizations to provide high-quality care that is more accessible, coordinated, and efficient, and that would ultimately improve patient centered outcomes. Using a Hybrid Type 1 effectiveness-implementation design will also allow us to assess contextual factors affecting widespread implementation and sustainment of each delivery modality.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18 inclusive
* Primary or co-primary DSM-V diagnosis of anxiety or OCD
* Symptom duration of at least 3 months
* Outpatient care needed
* Presence of a stable parent, or guardian, who can participate in treatment

Exclusion Criteria:

* Other primary or co-primary psychiatric disorder which requires initiation of other active current treatment
* Acute suicidality
* Concurrent psychotherapy
* Chronic medical illness that would preclude their active participation in treatment
* Treatment with psychotropic medication that is not stable

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 501 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale Second Edition: (CY-BOCS II) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The CY-BOCS II is a measure of obsessive-compulsive symptoms and their severity. The Obsession Rating Scale assesses five domains of obsessional severity, each scored from 0 (no impairment) to 5 (extreme impairment). The Compulsion Rating Scale assesses five domains of compulsion severity using the same 0-5 scale. The total OCD severity score ranges from 0 to 50, with higher scores indicating greater symptom severity.
Client Satisfaction Questionnaire-Revised (CSQ-8-R) | Week 8, Week 16 and follow-up (6 & 12 months)
  The CSQ-8-R measures consumer satisfaction with mental health services; satisfaction is measured using 8 items on a scale from 1 (Poor) to 4 (Excellent). Total satisfaction ranges from 8-32, with a high score indicating greater satisfaction.
Exposure Guide | Weekly at Week 1 through 24.
  The Exposure Guide is an empirically-supported exposure therapy fidelity/quality tool completed by study therapists. It measures exposure quality, including: therapist use of specific strategies that predict clinical improvement, exposure completion, exposure difficulty, therapeutic learning, barriers to completion, and engagement.
Pediatric Anxiety Rating Scale (PARS) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The PARS is a measure of anxiety symptoms and severity. The Anxiety Severity Items are 7 questions meant to assess the frequency of anxiety symptoms and associated impairment. Items are measured on a scale from 0 (none) to 5 (extreme).The total range of anxiety severity is reported on a scale from 0-35, with a higher score indicating greater severity.
Clinical Global Impression Scales | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The CGI is a clinician-rated measures of global severity and improvement. The Severity of illness scale reports the severity of current symptoms on a scale from 1 (not at all ill) to 7 (among the most extremely ill patients.) The Global Improvement Scale tracks improvement since treatment initiation on a scale from 1 (very much improved) to 7 (very much worse). The highest possible score on either scale is 7, indicating extreme severity or worse treatment outcome.
Top Problems Assessment | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The TPA is designed to independently solicit from youth and parents the top 3 problems they feel are most important to address in treatment. This is an idiographic measure of impairment that is driven by the individual needs and desires of the consumer. Respondents rate how much each problem bothers them from 0 ("not at all") to 10 (very, very much).
Child Sheehan Disability Scale (CSDS) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The CSDS measures the extent to which anxiety symptoms interfere with functioning. The Disability Scale measures the degree to which anxiety impacts school, social, and home life on a scale from 0 (Not at all) to 10 (very, very much.) Total anxiety-related impairment ranges from 0-30, with higher scores indicating greater impairment.
Barriers to Treatment Questionnaire - Parent Version (BTQ-P) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The BTQ-P is a 28-item measure adapted from the BTQ to assess parent perceptions of barriers to accessing treatment for their child's anxiety. The measure is completed at the outset of treatment and assesses such domains as logistic and financial barriers, stigma, and aspects of treatment. Items are rated on a 0 ("not at all true") to 2 ("mostly true") scale.

SECONDARY OUTCOMES:
Homework Compliance Form | Weekly at Week 1 though 24
  The measure tracks both the quality and quantity of homework completed between treatment sessions. This form has been used previously by our research group in large-scale treatment trials, and has been helpful in determining barriers to homework completion.
Demographics | Baseline
  We will assess participant demographics, including age, gender, sex assigned at birth, sexual orientation, race, and ethnicity. We will also assess perceived financial and food insecurity.
Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive and related Neuropsychiatric Disorders (DIAMOND-Kid) | Baseline
  DIAMOND-Kid is a brief, semi-structured diagnostic interview for DSM-5 psychiatric disorders in children and youth.
Caregiver Strain Questionnaire (CSQ) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The CSQ assesses parent perceptions of the extent to which caring for a child with emotional problems affects several domains, including family life and relationships, demands on time, financial strain, disruption of social life, worry, guilt, and fatigue. This is a 21-item self-report measure that calls for parents to rate the extent of strain for each item using a 0 ("not at all") to 4 ("very much") scale.
Reasons for Treatment Discontinuation form | Administered only at discharge, up to 6-months into study
  This is a case record form that documents any change in patient status (e.g., drop-out and premature termination) and the reasons for such changes.
Pediatric Accommodation Scale-Parent Report (PAS-PR) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  The PAS-PR is a 5-item questionnaire assessing the frequency and interference associated with accommodating the child's anxiety. Each item is followed by a series of common examples to illustrate the principle of accommodation for parents. Responses for frequency include 0 (never), 1 (rarely), 2 (occasionally), 3 (often), and 4 (always). Response options for interference due to accommodation include 0 (none), 1 (mild), 2 (moderate), 3 (severe), and 4 (extreme).
Ask Suicide Screening Questions (ASQ) | Baseline, Week 8, Week 16 and follow-up (6 & 12 months)
  ASQ assesses new or worsening suicidal ideation (SI) using four screening questions; a "yes" response to one or more items identifies 97% of youth at risk for suicide.
The Cultural Formulation Interview (CFI) | Baseline
  CFI supplements the diagnostic interview, gathering clinically relevant information about patient/family identities, perspectives of concerns, experiences with seeking mental health treatment, and sources of support
Everyday Discrimination Scale (EDS) | Baseline
  EDS measures perceived discrimination based on race and/or ethnicity.
Randomization Debrief | Administered at baseline
  We will record reactions from caregivers and child to treatment assignment using this clinician-rated measure. It includes capturing both verbatim responses from caregivers and child, as well as asking for interviewer impressions reactions from caregivers and child to treatment group assignment following randomization. The clinician also records the likelihood that the family will remain in the study and adhere to study protocols.
Treatment Expectancy | Administered at baseline
  This measure is a 3-item self-report questionnaire that captures parental beliefs about the efficacy about each treatment condition (In-person, telehealth, or flexible) using a scale from 1:"I expect my child will be very much improved," to 7: "I expect my child will be very much worse." The parent is also asked to select which treatment option would be best for their family. There is also a patient version of this measure used to capture patient beliefs about the efficacy about each treatment condition (in-person, virtual, or flexible) using the same scale. The patient is asked to select which treatment option they believe would be best for them and their family. The patient version of this measure will be completed by youth 12+.
End of Treatment Form | Administered only at discharge, up to 6-months into study
  This form captures whether the patient ended treatment before or at 6 months, as well as the reasons for discontinuation (e.g., scheduling, transportation, financial, treatment fit, symptoms) that apply. This form also gathers information about whether referrals were provided to the family upon study discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided